CLINICAL TRIAL: NCT06332001
Title: Evaluation of a Music and Interaction Intervention on Patient Distress During Whole Body Magnetic Resonance
Status: Recruiting | Type: Observational
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: IEO 1403
Record Dates: First submitted 2024-03-18; First posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Neoplasm Malignant
MeSH Terms: conditions — Neoplasms | interventions — Control Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental Group: Patients in this group receive the music and interaction interventions
  Interventions: Other: Experimental Group
- Control Group: Patients in this group receive a standard care condition (no music)
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Experimental Group — Listening of music of patient's choice during WB-MRI
  Groups: Experimental Group
Other: Control Group — Standard care condition during WB-MRI
  Groups: Control Group

SUMMARY:
This is a randomized controlled trial for the evaluation of the acceptability of Whole-Body-Magnetic Resonance Imaging (WB-MRI) based on music and comunication intervention compared to a standard care condition.

Subjects will be randomized into two groups: the experimental group or arm that receives the music and interaction interventions, and the control group or arm that receives a standard care condition.

DETAILED DESCRIPTION:
This study is a randomized controlled trial. Subjects referring to the European Institute of Oncology (IEO) and will undergo to WB-MRI for detection, staging, therapy monitoring or screening, will be asked to participate to the study and signed the informed consent.

Subjects will be divide into two groups: the experimental group or arm that receives the music and interaction interventions, and the control group or arm that receives a standard care condition.

The experimental group before the WB-MRI examination, complete distress Thermometer and received verbal information about the procedure from one of TRSM trained, during the examination subjects he has the opportunity to listen to the music of his choice and TRSM interacts with the subject four times to know he feels well. Before the examination control group complete distress Thermometer.

After examination both groups will be asked to complete a different WB-MRI acceptability questionnaire and distress Thermometer.

WB-MRI acceptability questionnaire is ad hoc questionnaire create to evaluate the acceptability of the WB-MRI based on of the interventions carried out.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who will undergo to WB-MRI for detection, staging, therapy monitoring or screening.
* Acceptance and signature of informed consent.

Exclusion Criteria:

* Any contra-indication to MRI examination (for example, pacemaker, in the first trimester of pregnancy, metal implants, etc.).
* Anxiety disorder and psychological or pharmacological treatments for anxiety

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects refferring to the European Institute of Oncology (IEO) and will undergo to WB-MRI for detection, staging, therapy monitoring or screening
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-12-31 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Acceptability of WB-MRI based on music and comunication intervention compared to a standard care condition. | 1 week
  Acceptability of WB-MRI based on music and comunication intervention compared to a standard care condition.
  The evaluation of the acceptability of WB-MRI will be done in both groups using an ad hoc WB-MRI acceptability questionnaire created to evaluate the acceptability of the WB-MRI based on of the interventions carried out

SECONDARY OUTCOMES:
Measure the level of patient's distress pre and post WB-MRI in the two groups using Distress Thermometer (V2.2020) | 1 week
  Patients randomized in both groups will complete Distress Thermometer (Version 2.2020) to assess the level of distress before and after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Petralia, Principal Investigator — European Institute of Oncology
Locations (1):
- IEO Istituto Europeo di Oncologia, Milan, Italy